CLINICAL TRIAL: NCT05368545
Title: Influence of Intensive Lipid-lowering Witgh Statin and Ezetimibe Prescription on Computed Tomography Derived Fractional Flow Reserve in Patients With Stable Chest Pain
Brief Title: Influence of Lipid Lowering on Impaired Coronary Flow
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aarhus University Hospital (Other)
Collaborators: HeartFlow, Inc. (Industry)
Responsible Party: Principal Investigator, Bjarne Linde Nørgaard, Professor, MD, DMSc, PhD, Aarhus University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: AahusUH; 2019-001912-50 (EudraCT Number)
Record Dates: First submitted 2022-05-06; First posted 2022-05-10 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2025-04

CONDITIONS: Coronary Artery Disease
Keywords: fractional flow reserve; CT derived fractional flow reserve; coronary artery disease; ischemic heart disease; stable chest pain; statin; blood cholesterol level
MeSH Terms: conditions — Coronary Artery Disease; Myocardial Ischemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- usual care lipid lowering (Active Comparator): Usual care: atorvastatin 40 mg
  Interventions: Drug: High intensity lipid lowering
- Intensive lipid lowering (Experimental): Intensive: rosuvastatin 40 mg + ezetimibe 10 mg
  Interventions: Drug: High intensity lipid lowering

INTERVENTIONS:
Drug: High intensity lipid lowering — Two different regimens of drugs with different effects on LDL lowering
  Other Names: Usual care lipid lowering

SUMMARY:
This study assess in patients with stable chest pain and coronary artery disease (CAD) determined by coronary CTA whether cholesterol lowering with regression of coronary adverse plaque characteristics is associated with recovery of impaired flow

DETAILED DESCRIPTION:
Multicenter, prospective study. 105 patients with stable chest pain, and moderate CAD, statin naive (and LDL cholesterol >2 mM), and at least one translesional FFRct value <0.81 are randomized (patients with significant CAD in the left main or other proximal segments are excluded from the study) to either "atorvastatin 40 mg daily" or "rosuvastatin 40 mg + ezetimibe 10 mg daily" treatment. Patients are followed for 18 months with 2 CT scans performed at 9 months and one at 18 months. At each 4 CT scans blinded corelab analyses of plaque characteristics and volumes as well as FFRct calculation (HeartFlow) are performed. The primary endpoint is changes in FFRct values from 0 to 18 months. Secondary endpoints are 1 changes in FFRct values from 0 to 9 months of follow-up, and changes in low density plaques volumes and number of lesions with positive remodeling over time relative to changes in LDL cholesterol.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥35 y
* Symptoms suggestive of stable CAD
* No pre-CTA known CAD
* At least one lesion with FFRct <0.81
* Sinus rhythm
* LDL cholesterol >2.0 mM
* Statin use >2 months
* Life expentancy < 3 years
* Signed informed consent

Exclusion Criteria:

* Known CAD
* Poor CTA image quality inadequiate for FFRct analysis (determined by corelab)
* Significant CAD in the left main or proximal coronary segments
* Referral to invasive catheterization
* Statin intolerance
* BMI >40
* Allergy to ionidated contrast
* Pregnancy

Min Age: 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 109 (Actual)
Dates: Start 2020-05-15 (Actual); Primary Completion 2024-04-17 (Actual); Study Completion 2024-04-17 (Actual)

PRIMARY OUTCOMES:
Changes in FFRct values | 18 months
  CT derived FFR

SECONDARY OUTCOMES:
Changes in FFRct values | 9 months
  CT derived FFR
Changes in low density plaque volumes | 0-9, and 0-18 months
  CT determined plaque volumes

CONTACTS AND LOCATIONS:
Overall Officials: Bjarne Norgaard, MD, PhD, Principal Investigator — Aarhus University Hospital
Locations (1):
- Aarhus University Hospital, Aarhus, Denamrk, Denmark

IPD SHARING:
Plan to Share IPD: No